CLINICAL TRIAL: NCT01438307
Title: Phase II Study of a Novel Taxane (Cabazitaxel-XRP6258) in Previously Treated Advanced Non-Small Cell Lung Cancer (NSCLC) Patients
Brief Title: Phase II Study of Cabazitaxel-XRP6258 in Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Francisco Robert,MD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F110512012 (UAB 1021); UAB 1021 (Other: institutional study identifier number)
Record Dates: First submitted 2011-09-15; First posted 2011-09-22 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Stage IV NSCLC; Metastatic NSCLC
Keywords: Non-small cell lung cancer; Cabazitaxel-XRP6258; P-glycoprotein; taxane; Advanced NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Schedule A (Experimental): Subjects with advanced non-small cell lung cancer who have been previously treated will be given a specific regimen of the novel taxane, Cabazitaxel-XRP6258.
  Subjects with asymptomatic brain metastases will be eligible for the study and a subset analysis will take place to help determine what, if any, effect Cabazitaxel-XRP6258 has on brain metastases.
  Interventions: Drug: Cabazitaxel-XRP6258 (3-week cycle)
- Schedule B (Experimental): Subjects with advanced non-small cell lung cancer who have been previously treated will be given a specific regimen of the novel taxane, Cabazitaxel-XRP6258, different from Schedule A.
  Subjects with asymptomatic brain metastases will be eligible for the study and a subset analysis will take place to help determine what, if any, effect Cabazitaxel-XRP6258 has on brain metastases.
  Interventions: Drug: Cabazitaxel-XRP6258 (5-week cycle)

INTERVENTIONS:
Drug: Cabazitaxel-XRP6258 (3-week cycle) — Subjects in Schedule A will begin with an initial dose of 20 mg/m2 every 3 weeks as a 1 hour IV infusion. If no dose limiting toxicities are experienced after cycle 1, then the dose will be escalated to 25 mg/m2. Treatment with Cabazitaxel-XRP6258 will continue for a total of 6 cycles unless there is evidence of disease progression, intolerable toxicity or withdrawal of consent. Further treatment after 6 cycles of treatment in patients who achieved an objective response or stable disease, and no significant toxicity will be an individual decision from the investigator.
  Other Names: Jevtana
  Arms: Schedule A
Drug: Cabazitaxel-XRP6258 (5-week cycle) — Subjects in Schedule B will begin with an initial dose of 8.4 mg/m2 as a 1 hour IV infusion on days 1, 8, 15, and 22 of a 5-week cycle. If no dose limiting toxicities are experienced after cycle 1, then the dose will be escalated to 10 mg/m2. Treatment with Cabazitaxel-XRP6258 will continue for a total of 6 cycles unless there is evidence of disease progression, intolerable toxicity or withdrawal of consent. Further treatment after 6 cycles of treatment in patients who achieved an objective response or stable disease, and no significant toxicity will be an individual decision from the investigator.
  Other Names: Jevtana
  Arms: Schedule B

SUMMARY:
Lung cancer is the leading cause of cancer death worldwide and in the United States. The majority of lung cancers are non-small cell lung cancer (NSCLC). The majority of NSCLC cases are advanced at the time of diagnosis. Chemotherapy has improved overall survival but remains limited at < 12 months median overall survival. New approaches are needed for second line chemotherapy treatment. Cabazitaxel-XRP6258 has shown increased overall survival in metastatic prostate cancer and it is hopeful it can do the same in advanced NSCLC.

DETAILED DESCRIPTION:
A substantial number of patients with lung cancer progress after first line treatment and require second line chemotherapy. Lung cancer appears to account for 40-50% of all known brain metastasis. The incidence of brain metastases among lung cancer patients ranges from 16-20%. Chemotherapy has had limited utility due to problems crossing the blood brain barrier.

Currently there are three drugs approved by the FDA for second line treatment of NSCLC but each has distinct toxicities. Cabazitaxel-XRP6258 is a potent novel taxane with enhanced activity against an increased number of cell lines including lung, prostate, colon, pancreas, head and neck, kidney, gastric, glioblastoma, and melanoma. It also has the ability to cross the blood brain barrier. Cabazitaxel-XRP6258 was found to have an improved antiproliferative activity than other chemotherapy agents against insensitive cell lines. The Phase I studies of Cabazitaxel-SRP6258 have determined dosage and schedule recommendations in advanced NSCLC patients to be utilized for a Phase II multicenter study.

Subjects will be placed on one of two schedules (A or B) each with a specified dosage and administration schedule. All subjects will be followed for survival/progression after every 2 cycles of therapy with imaging studies. A two stage design will be used for each of the two schedules. Fourteen subjects will be accrued for each schedule in the first stage with possible accrual of an additional 34 subjects per schedule depending upon the first stage results.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of NSCLC (squamous or non-squamous or NSCLC-not specified)
* Subjects who have failed first line chemotherapy (platinum doublets or non- platinum doublets [previous taxane exposure is allowed]) for Stage IV NSCLC.
* Measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Age > 18 years old
* Adequate bone marrow, liver and renal function, defined as:

  * Absolute neutrophil count (ANC) greater than or equal to 1500/ul
  * Hemoglobin greater than or equal to 10 g/dl
  * Platelet count greater than or equal to 100,000/ul
  * Total bilirubin less than or equal to 1.5 x upper limit of normal (except in subjects with documented Gilbert's syndrome)
  * AST/ALT less than or equal to 1.5 x upper limit of normal
  * Serum creatinine less than or equal to 1.8 mg/dl
* Fully recovered from any previous surgery (at least 4 weeks since major surgery)
* Fully recovered from previous radiation therapy (at least 2 weeks)
* All subjects must agree to practice approved methods of birth control (if applicable). A negative pregnancy test must be documented during the screening period for women of childbearing potential.
* Written informed consent and authorization to use and disclose health information (HIPAA) must be signed by the subject.
* Subjects with symptomatic brain metastases should be adequately treated and controlled prior to the initiation of the study. Subjects with asymptomatic brain metastases will be allowed in the study without any prior therapy for brain metastases.

Exclusion Criteria:

* Concurrent cancer chemotherapy, biologic therapy or radiotherapy
* Administration of any investigational agent within 28 days prior to administration of current therapy
* Untreated symptomatic brain metastases
* Greater than or equal to Grade 2 neuropathy
* Concurrent serious infection
* Concomitant severe or uncontrolled underlying medical disease unrelated to the tumor, which is likely to compromise subject safety and affect the outcome of the study.
* Treatment for a cancer other the NSCLC within 5 years prior to enrollment, with the exception of basal cell carcinoma or carcinoma in situ of the cervix
* Any evidence of history of hypersensitivity for the taxane class of chemotherapy drugs
* History of positive serology for HIV
* Psychiatric disorder that prevents subjects from providing informed consent or following protocol instructions
* Pregnant or lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Georgia Cancer Center, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be randomized to one of two schedules (A or B) each with a specified dosage and administration schedule. A two stage design will be used for each of the two schedules. Fourteen subjects will be accrued for each schedule in Stage I with an additional 34 subjects in Stage II per schedule depending upon the first stage results.
Pre-assignment Details: New approaches are needed for 2nd line chemotherapy treatment. Cabazitaxel-XRP6258 has shown increased overall survival in metastatic prostate cancer and it is hopeful to do the same in advanced Non-Small Cell Lung Cancer (NSCLC).This phase II study will evaluate the efficacy of cabazitaxel chemotherapy in 2nd line setting in patients with NSCLC.
Groups:
- Treatment Schedule A: Cabazitaxel 20 mg/m2 every 3 weeks as a 1 hour IV infusion with a planned dose escalation of to 25 mg/m2 if no dose limiting toxicities (DLTs) were observed.
  All subjects will be followed for survival/progression after every 2 cycles of therapy with imaging studies.
- Treatment Schedule B: Cabazitaxel 8.4 mg/m2 weekly on Days 1, 85, 15, and 22 of a 5 week cycle with a planned dose escalation to 10 mg/m2 weekly if no dose limiting toxicities (DLTs) were observed.
  All subjects will be followed for survival/progression after every 2 cycles of therapy with imaging studies.
Period: Overall Study
Arm/Group | Treatment Schedule A | Treatment Schedule B
Started | 14 | 14
Completed | 13 | 13
Not Completed | 1 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Schedule A: Cabazitaxel 20 mg/m2 every 3 weeks as a 1 hour IV infusion with a planned dose escalation of to 25 mg/m2 if no dose limiting toxicities (DLTs) were observed.
- Schedule B: Cabazitaxel 8.4 mg/m2 weekly on Days 1, 85, 15, and 22 of a 5 week cycle with a planned dose escalation to 10 mg/m2 weekly if no dose limiting toxicities (DLTs) were observed.
- Total: Total of all reporting groups
Arm/Group | Schedule A | Schedule B | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 15
  >=65 years | 9 | 4 | 13
Age, Continuous [Median (Full Range); unit: Years] | 68 [47 to 79] | 64 [41 to 78] | 65 [41 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The objective response is defined as the percentage of patients that achieve a complete and/or partial response according to The Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1).
Time Frame: Baseline up to 28 months
Measure: Number; unit: participants
Groups:
- Schedule A: Subjects with advanced non-small cell lung cancer who have been previously treated will be given a specific regimen of the novel taxane, Cabazitaxel-XRP6258.
  Subjects with asymptomatic brain metastases will be eligible for the study and a subset analysis will take place to help determine what, if any, effect Cabazitaxel-XRP6258 has on brain metastases.
  Cabazitaxel-XRP6258 (3-week cycle): Subjects in Schedule A will begin with an initial dose of 20 mg/m2 every 3 weeks as a 1 hour IV infusion. If no dose limiting toxicities are experienced after cycle 1, then the dose will be escalated to 25 mg/m2. Treatment with Cabazitaxel-XRP6258 will continue for a total of 6 cycles unless there is evidence of disease progression, intolerable toxicity or withdrawal of consent. Further treatment after 6 cycles of treatment in patients who achieved an objective response or stable disease, and no significant toxicity will be an individual decision from the investigator.
- Schedule B: Subjects with advanced NSCLC who have been previously treated will be given a specific regimen of the novel taxane, Cabazitaxel-XRP6258, different from Schedule A.
  Subjects with asymptomatic brain metastases will be eligible for the study and a subset analysis will take place to help determine what, if any, effect Cabazitaxel-XRP6258 has on brain metastases.
  Cabazitaxel-XRP6258 (5-week cycle): Subjects in Schedule B will begin with an initial dose of 8.4 mg/m2 as a 1 hour IV infusion on days 1, 8, 15, and 22 of a 5-week cycle. If no dose limiting toxicities are experienced after cycle 1, then the dose will be escalated to 10 mg/m2. Treatment with Cabazitaxel-XRP6258 will continue for a total of 6 cycles unless there is evidence of disease progression, intolerable toxicity or withdrawal of consent. Further treatment after 6 cycles of treatment in patients who achieved an objective response or stable disease, and no significant toxicity will be an individual de
Arm/Group | Schedule A | Schedule B
Number analyzed (Participants) | 13 | 13
participants | 0 | 1

2. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival is defined from the initiation of treatment until radiological-clinical evidence of progression according to the RECIST (v 1.1).
Time Frame: Baseline up to 28 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Schedule A | Schedule B
Number analyzed (Participants) | 13 | 13
months | 3 [1.0 to 5.0] | 3 [2.0 to 3.0]

3. Secondary Outcome: Number of Patients With Any Graded Adverse Event
Description: Safety will be assessed using the National Cancer Institute Common Toxicity Criteria (Version 4.0) and all adverse events will be recorded prior to each treatment regimen.
Time Frame: Baseline up to 28 months
Population: 14 patients in each cohort were included in the toxicity assessment and 13 patients in each cohort in the efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule A | Schedule B
Number analyzed (Participants) | 14 | 14
Participants | 14 | 14

4. Secondary Outcome: Overall Survival
Description: Assessment will be made in subjects with Stage IV NSCLC who receive Cabazitaxel-SRP6258 after progressing with first line platinum-based chemotherapy.
Time Frame: 28 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Schedule A | Schedule B
Number analyzed (Participants) | 13 | 13
months | 6 [0.50 to 7.0] | 13 [0.50 to 14.0]

ADVERSE EVENTS:
Time Frame: 28 Months
Arm/Group | Treatment Schedule A | Treatment Schedule B
All-Cause Mortality (participants affected / at risk) | 1/14 | 1/14
Serious Adverse Events (participants affected / at risk) | 7/14 | 1/14
Other Adverse Events (participants affected / at risk) | 5/14 | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Schedule A (N=14) | Treatment Schedule B (N=14)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 0 (0) — 6 patients from Schedule A experience neutropenia (grade =/>3).
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Schedule A (N=14) | Treatment Schedule B (N=14)
Neuropathy (Nervous system disorders) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No